CLINICAL TRIAL: NCT02768493
Title: Ultrasonographic Assessment of Optic Nerve Sheath Diameter in Children Receiving Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4-2016-0192
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Orchiopexy; Inguinal Hernioplasty; Hydrocelectomy; Diverticulectomy; Fistula Repair; Penoplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low dose group (Experimental): Patients in the low dose group are given 1.0 ml/kg of 0.15% ropivacaine for caudal block.
  Interventions: Drug: 1.0 ml/kg of 0.15% ropivacaine
- high dose group (Active Comparator): Patients in the high dose group are given 1.5 ml/kg of 0.15% ropivacaine for caudal block.
  Interventions: Drug: 1.5 ml/kg of 0.15% ropivacaine

INTERVENTIONS:
Drug: 1.0 ml/kg of 0.15% ropivacaine — Randomly selected patients of the high dose group are given 1.5 ml/kg of 0.15% ropivacaine for caudal block before their surgery. In contrast, patients in the low dose group are given 1.0 ml/kg of 0.15% ropivacaine for caudal block before surgery.
  Arms: low dose group
Drug: 1.5 ml/kg of 0.15% ropivacaine — Randomly selected patients of the high dose group are given 1.5 ml/kg of 0.15% ropivacaine for caudal block before their surgery. In contrast, patients in the low dose group are given 1.0 ml/kg of 0.15% ropivacaine for caudal block before surgery.
  Arms: high dose group

SUMMARY:
The recent study revealed that high-volume caudal block caused reduction in cerebral blood flow velocity and cerebral oxygenation. It was supposed to be associated with increased intracranial pressure. Ultrasonography of optic nerve sheath diameter shows a good level of diagnostic accuracy for detecting intracranial hypertension. The aim of this study is to evaluate the effect of caudal block on intracranial pressure in pediatric patients undergoing urologic surgery. Eighty patients, aged 6 months to 4 years, receiving caudal block before urologic surgery will be divided into high dose group (n=40) and low dose group (n=40). Randomly selected patients of the high dose group are given 1.5 ml/kg of 0.15% ropivacaine for caudal block. In contrast, patients in the low dose group are given 1.0 ml/kg of 0.15% ropivacaine for caudal block. The primary endpoint is the optic nerve sheath diameter after caudal block measured by optic nerve ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients
* weighing less than 16 kg
* who receive caudal block before urologic surgery

Exclusion Criteria:

* Subjects are ineligible if they have contraindication for caudal block such as infection, coagulopathy, anomaly, or past medical history related to increased intracranial pressure
* ophthalmic disease
* expected operation time is less than 30 minutes
* both parents are unable to communicate or speak Korean.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The difference in the optic nerve sheath diameter between groups | 1 day

SECONDARY OUTCOMES:
The variation in the optic nerve sheath diameter before and after caudal block | 30 minutes
the difference in the variation of the optic nerve sheath diameter between groups | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei universiy college of medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girisgin AS, Kalkan E, Kocak S, Cander B, Gul M, Semiz M. The role of optic nerve ultrasonography in the diagnosis of elevated intracranial pressure. Emerg Med J. 2007 Apr;24(4):251-4. doi: 10.1136/emj.2006.040931. PMID 17384377
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019
- [Background] Lundblad M, Forestier J, Marhofer D, Eksborg S, Winberg P, Lonnqvist PA. Reduction of cerebral mean blood flow velocity and oxygenation after high-volume (1.5 ml kg(-)(1)) caudal block in infants. Br J Anaesth. 2014 Oct;113(4):688-94. doi: 10.1093/bja/aeu161. Epub 2014 Jun 27. PMID 24972788
- [Derived] Lee B, Koo BN, Choi YS, Kil HK, Kim MS, Lee JH. Effect of caudal block using different volumes of local anaesthetic on optic nerve sheath diameter in children: a prospective, randomized trial. Br J Anaesth. 2017 May 1;118(5):781-787. doi: 10.1093/bja/aex078. PMID 28486629